CLINICAL TRIAL: NCT05388370
Title: Post-Authorisation Safety Study of Paediatric Patients Initiating Selumetinib: A Multiple-Country Prospective Cohort Study.
Brief Title: PASS of Paediatric Patients Initiating Selumetinib
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1346R00004
Record Dates: First submitted 2022-04-12; First posted 2022-05-24 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Neurofibromatosis Type 1
MeSH Terms: conditions — Neurofibromatosis 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Base Cohort: The Base Cohort includes all enrolled patients aged 3 to < 18 years.
- Nested Prospective Cohort: The Nested Prospective Cohort will include the subset of Base Cohort patients aged 8 to < 18 years who have not reached Tanner Stage V on the index date

SUMMARY:
Neurofibromatosis type 1 (NF1) is a rare, autosomal dominant genetic disorder that is caused by germline mutations in the NF1 tumour suppressor gene, which encodes the tumour suppressor protein neurofibromin 1. Plexiform neurofibromas (PN) are histologically benign nerve sheath tumours, which typically grow along large nerves and plexi.

On 5 March 2020, a centralised Marketing Authorisation Application was submitted to the European Medicines Agency (EMA), Marketing Authorisation in EU was granted on 17 Jun 2021.

As part of the approval process, a Risk Management Plan (RMP) was developed and submitted to the EMA to summarise the safety concerns emerging from the clinical development program. The RMP included additional pharmacovigilance plans for a noninterventional Post-authorisation Safety Study (PASS) to further characterise the safety of selumetinib in paediatric patients with NF1-related PN in routine clinical practice.

The planned non-interventional PASS will address gaps in knowledge identified by the RMP, including the important identified risk and some of the potential risks and missing information on long-term developmental toxicity in children, by characterising the safety profile associated with selumetinib use among paediatric patients (age d 8 to < 18 years old) with a diagnosis of NF1 with symptomatic, inoperable PN.

This study is a specific obligation in the context of a conditional marketing authorisation for selumetinib (ie, Category 2 PASS). Study results will contribute to updating the safety profile of selumetinib in a relatively large population of patients with different personal characteristics across multiple health care systems and patterns of real-world clinical practice in European countries and Israel.

The study will enrol 2 cohorts:

1. The Base Cohort includes all enrolled patients aged 3 to < 18 years.
2. The Nested Prospective Cohort will include the subset of Base Cohort patients aged 8 to < 18 years who have not reached Tanner Stage V on the index date.

DETAILED DESCRIPTION:
Neurofibromatosis type 1 (NF1) is a rare, autosomal dominant genetic disorder that is caused by germline mutations in the NF1 tumour suppressor gene, which encodes the tumour suppressor protein neurofibromin 1. Plexiform neurofibromas (PN) are histologically benign nerve sheath tumours, which typically grow along large nerves and plexi.

On 5 March 2020, a centralized Marketing Authorisation Application was submitted to the European Medicines Agency (EMA), Marketing Authorization in EU was granted on 17 Jun 2021.

As part of the approval process, a Risk Management Plan (RMP) was developed and submitted to the EMA to summarise the safety concerns emerging from the clinical development program. The RMP included additional pharmacovigilance plans for a non-interventional Post-authorisation Safety Study (PASS) to further characterise the safety of selumetinib in paediatric patients with NF1-related PN in routine clinical practice.

The RMP version 1.0 (succession 4) approved by EMA on 22 April 2021 had 1 important identified risk with selumetinib treatment:

-LVEF reduction

The RMP also identified 5 important potential risks with selumetinib treatment:

* Physeal dysplasia
* Ocular toxicity
* Myopathy
* Hepatotoxicity
* Choking on the capsule Long-term exposure (including long-term safety data on developmental toxicity in children) was identified in the RMP as an area of missing information.

The planned non-interventional PASS will address gaps in knowledge identified by the RMP, including the important identified risk and some of the potential risks and missing information on long-term developmental toxicity in children, by characterising the safety profile associated with selumetinib use among paediatric patients (aged d 8 to < 18 years old) with a diagnosis of NF1 with symptomatic, inoperable PN.

This study is a specific obligation in the context of a conditional marketing authorisation for selumetinib (ie, Category 2 PASS). Study results will contribute to updating the safety profile of selumetinib in a relatively large population of patients with different personal characteristics across multiple health care systems and patterns of real-world clinical practice in up to 52 specialist clinics for the treatment of pediatric patients with NF1 across up to 12 European countries and in Israel.

The primary objective of this study is:

- To characterise the safety of selumetinib, including up to 6 years of long-term safety, in paediatric patients with NF1-related symptomatic, inoperable PN, 8 to < 18 years old who have not reached Tanner Stage V at the start of selumetinib treatment (Nested Prospective Cohort).

The secondary objective of this study is:

- To describe the demographic and clinical profile of the paediatric population 3 to < 18 years old with NF1-related symptomatic inoperable PN who start selumetinib in routine clinical practice (Base Cohort).

The study observation period was anticipated to begin in Q2 of 2022, with some variation by country (actual start date was 23 May 2022). Patients will be enrolled after selumetinib access is commercially available and patients are able to receive the medicine as part of local clinical practice.

The target population for this study are patients with NF1 in the EU with symptomatic, inoperable PN who have been prescribed at least 1 dose of selumetinib and who are aged 3 to < 18 years at the start of selumetinib treatment, except for those patients receiving treatment with a mitogen-activated protein kinase inhibitor before the index date.

The study will enrol 2 cohorts:

1. The Base Cohort includes all enrolled patients aged 3 to < 18 years.
2. The Nested Prospective Cohort will include the subset of Base Cohort patients aged 8 to < 18 years who have not reached Tanner Stage V on the index date.

Patient screening will be conducted throughout the enrolment period and baseline data for all patients will be abstracted from medical records. Those meeting the criteria for enrolment in the Nested Prospective Cohort will be followed up during their routine standard of care visits with the treating clinician (expected to occur every 6 to 12 months) for up to 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with NF1 with symptomatic, inoperable PN
* Have initial treatment with selumetinib up to 6 months (i.e.182 days)prior to enrolment into the study (i.e. signature of the ICF)
* Are aged 3 years and above, and are < 18 years of age on the index date
* Parent or legal guardian, as required by country-specific regulation, have provided informed consent (unless a country-specific waiver is obtained) Additional Criteria for Nested Prospective Cohort
* Are at least 8 years old and
* Are prior to attainment of Tanner Stage V on the index date

Exclusion Criteria:

* Have received treatment with a mitogen-activated protein kinase inhibitor before the index date
* Are participating in an interventional study at index date

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The target population for this study are patients with NF1 with symptomatic, inoperable PN who have been prescribed at least 1 dose of selumetinib and who are aged 3 to < 18 years at the start of selumetinib treatment, except for those patients receiving treatment with a mitogen-activated protein kinase inhibitor before the index date.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2028-05-23 (Estimated); Study Completion 2028-05-23 (Estimated)

PRIMARY OUTCOMES:
LVEF reduction | at routine clinical care throughout the follow up, with frequency of 6 to 12 months
  LVEF reduction will be detected as present or absent and when present if symptomatic or asymptomatic. All cardiac tests conducted will be collected Measured on routine echocardiogram or a cardiac MRI (CT, angiography, etc.) and then collected into the study from the medical records.
Occurrence of Physeal dysplasia after treatment start | at routine clinical care throughout the follow up, with frequency of 6 to 12 months
  Physeal dysplasia will be detected as present or absent based on the physician reading of: MRI: Knee (preferred) or wrist X-ray: Knee (preferred) and/or wrist to assess growth plate Height and weight records
Rise of serum creatine phosphokinase levels AND concurrent musculoskeletal symptoms | at routine clinical care throughout the follow up, with frequency of 6 to 12 months, up to 6 years
  A clinically meaningful rise in serum creatine phosphokinase (eg, above the normal limit or increase by 1 or more CTCAE grade shift) combined with musculoskeletal symptoms will be detected as present or absent based on the physician's reading, as a marker of potential myopathy
Rise in transaminase (ALT and AST) and concurrent rise in bilirubin | at routine clinical care throughout the follow up, with frequency of 6 to 12 months, up to 6 years
  A clinically meaningful rise in the measured levels (eg, above the normal limit or increase by 1 or more CTCAE grade shift) will be detected as present or absent, and when present if symptomatic or asymptomatic, as a marker of potential hepatotoxicity
Cumulative incidence of ocular toxicity | at routine clinical care throughout the follow up, with frequency of 6 to 12 months
  An abnormal ocular examination will be detected as present or absent based on the physician's reading, as a marker of potential ocular toxicity
Cumulative incidence of Abnormal pubertal development | at routine clinical care throughout the follow up, with frequency of 6 to 12 months
  Tanner stage criteria (Stages I-V). Abnormal pubertal development will require interpretation by the Investigator with respect to Tanner Stage in the context of the patient's age; recorded as normal or abnormal (if abnormal, further specified as delayed puberty or precocious puberty)

SECONDARY OUTCOMES:
baseline data - demographics | At baseline - most recent assessments made within 365 days before the index date
  Demographics: Age
baseline data - demographics | At baseline - most recent assessments made within 365 days before the index date
  sex
baseline data - demographics | At baseline - most recent assessments made within 365 days before the index date
  height (cm)
baseline data - demographics | At baseline - most recent assessments made within 365 days before the index date
  weight (kg)
baseline data - demographics | At baseline - most recent assessments made within 365 days before the index date
  Tanner staging level
baseline data - demographics | At baseline - most recent assessments made within 365 days before the index date
  Ethnicity (where allowed by GDPR/privacy laws)
Baseline data - Clinical characteristics | At baseline - most recent assessments made within 365 days before the index date
  PN(s) (number, location, classification and morbidities)
Baseline data - Clinical characteristics | At baseline - most recent assessments made within 365 days before the index date
  prior medication and relevant procedures, concomitant medications
Baseline data - Clinical characteristics | At baseline - most recent assessments made within 365 days before the index date
  date of initial NF1 and PN diagnosis, NF1 origin (familial or spontaneous), and any genetic testing results

OTHER OUTCOMES:
Other Variables and Covariates | at baseline and throughout follow-up, up to 6 years
  Height (cm)
Other Variables and Covariates | at baseline and throughout follow-up, up to 6 years
  Weight (kg)
Other Variables and Covariates | at baseline and throughout follow-up, up to 6 years
  Body surface area
Other Variables and Covariates | at baseline and throughout follow-up, up to 6 years
  Tanner staging (level from I to V)
Other Variables and Covariates | at baseline and throughout follow-up, up to 6 years
  Concomitant medications, including any medications used to treat AEs
Other Variables and Covariates | at baseline and throughout follow-up, up to 6 years
  Comorbidities
Other Variables and Covariates | at baseline and throughout follow-up, up to 6 years
  NF1-related clinical manifestation and complications
Other Variables and Covariates | at baseline and throughout follow-up, up to 6 years
  PN-related variables (including for any clinically important target PNs)
Other Variables and Covariates | at baseline and throughout follow-up, up to 6 years
  PN-related symptoms/morbidities

CONTACTS AND LOCATIONS:
Locations (45):
- Research Site, Vienna, Austria
- France (12):
  - Research Site, Amiens
  - Research Site, Angers
  - Research Site, Bordeaux
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Rennes
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Villejuif
- Germany (5):
  - Research Site, Dresden
  - Research Site, Duisburg
  - Research Site, Hamburg
  - Research Site, München
  - Research Site, Tübingen
- Israel (3):
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Italy (8):
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Pavia
  - Research Site, Roma
  - Research Site, Torino
  - Research Site, Trieste
- Research Site, Rotterdam, Netherlands
- Portugal (2):
  - Research Site, Lisbon
  - Research Site, Porto
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Esplugues de Llobregat
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Santiago de Compostela
  - Research Site, Seville
- Switzerland (4):
  - Research Site, Basel
  - Research Site, Bern
  - Research Site, Lausanne
  - Research Site, Sankt Gallen
- United Kingdom (3):
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, study progress reports, and final study report will be included in regulatory communications in line with the RMP, PSUR, and other regulatory reporting requirements. Study reports will be prepared using a template following the GVP Module VIII Section B.6.3.
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Background] EMA2017b EMA. Guideline on good pharmacovigilance practices (GVP). Module VIII - Post-authorisation safety studies (EMA/813938/2011 Rev 3). European Medicines Agency; 09 October 2017b. Available at: https://www.ema.europa.eu/documents/scientificguideline/ guideline-good-pharmacovigilance-practices-gvp-
- [Background] International Committee Of Medical Journal Editors. [Recommendations for the conduct, reporting, editing and publication of scholarly work in medical journals (revised in January 2024): a Korean translation]. Ewha Med J. 2024 Oct;47(4):e48. doi: 10.12771/emj.2024.e48. Epub 2024 Oct 31. No abstract available. Korean. PMID 40704003
- [Background] ISPE. Guidelines for good pharmacoepidemiology practices (GPP). Pharmacoepidemiol Drug Saf. 2008 Feb;17(2):200-8. doi: 10.1002/pds.1471. No abstract available. PMID 17868186
- [Background] KOSELUGO (selumetinib) KOSELUGO (selumetinib) capsules, for oral use, initial US Approval: 2020. Distributed by: AstraZeneca Pharmaceuticals LP, Wilmington, DE 19850. USPI revised April 2020, Reference ID 4590044.
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. Lancet. 2007 Oct 20;370(9596):1453-7. doi: 10.1016/S0140-6736(07)61602-X. PMID 18064739